CLINICAL TRIAL: NCT00759044
Title: Validation of a New Methodology for Mapping the Human Blood-Retinal Barrier Function
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: CNTM023A
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Age-Related Maculopathy; Diabetic Macular Edema
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- AMD: Patients diagnosed with AMD
- DME: Patients diagnosed with DME

SUMMARY:
To validate a new methodology, named Retinal Leakage Analysis (RLA), for mapping the human Blood-Retinal Barrier (BRB) function, in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AMD, or
* Patients diagnosed with DME
* Age over 18 years
* Inform consent

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations
* Glaucoma
* Dilatation of the pupil < 5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with AMD or DME followed regularly by their ophthalmologist at the AIBILI Clinical Trial Center will be asked to perform additional optical examinations as a continuation of the routine fluorescein angiographies (FA).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Blood-Retinal Barrier (BRB) function measured by Retinal Leakage Analysis (RLA).

CONTACTS AND LOCATIONS:
Overall Officials: José G Cunha-Vaz, Prof., Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI Clinical Trial Center, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Background] Bernardes R, Dias J, Cunha-Vaz J. Mapping the human blood-retinal barrier function. IEEE Trans Biomed Eng. 2005 Jan;52(1):106-16. doi: 10.1109/TBME.2004.839801. PMID 15651569